CLINICAL TRIAL: NCT06347510
Title: Does the Level of ST2 in Pediatric Heart Failure Patients Indicate the Likelihood of Cardiovascular Events and Mortality?
Brief Title: The Level of sST2 in Pediatric Heart Failure
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ayse Sulu, Assistant Professor/ Pediatric Cardiology, Eskisehir Osmangazi University
Other Study IDs: E-25403353-050.99-174660
Record Dates: First submitted 2024-03-26; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Congenital Heart Disease; Congestive Heart Failure
Keywords: Suppression of tumorigenicity 2 (ST2); congenital heart disease; congestive heart failure
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Suppression of tumorigenicity 2 (ST2) — Suppression of tumorigenicity 2 (ST2) is a member of the interleukin-1 (IL-1) receptor family. The ligand and soluble versions are its two isoforms. It was first isolated in 1989. It was found to function as an IL-33 ligand in 2005. The IL-33-ST2L ligand complex's creation offers protection against heart fibrosis and hypertrophy. The formation of this complex is inhibited by soluble ST2, which removes the cardioprotective effect. Unlike NT pro BNP, it is unaffected by age, body mass index, creatinine, hemoglobin, and albumin levels, according to studies performed on individuals. with heart failure.

SUMMARY:
Introduction: Suppression of tumorigenicity 2 (ST2) is a receptor member belongs to the Interleukin-1 (IL-1) family. The ligand and soluble versions are its two isoforms. The interleukin-33-ST2 ligand complexs development provides protection against heart fibrosis and hypertrophy. Investigations on heart failure in adults has demonstrated that it does not change by age, body mass index (BMI), creatinine, hemoglobin, and albumin levels, in contrast to NT pro brain natriuretric peptit. In adult heart failure patients, it has been demonstrated to be an independent predictor of mortality and cardiovascular events. The most recent guideline recommends using it as class 2b in the diagnosis of adult heart failure. Studies on ST2 in children are rare. The purpose of this study is to assess the prognostic value of ST2 for cardiovascular events in young individuals suffering from heart failure.

Method: The study included pediatric patients (0-18 years old) with congenital heart disease or cardiomyopathy who needed medical care as well as surgical or interventional treatment. Height, weight, gender, saturation, heart failure classification (Ross or New York heart Assosiation), medications taken, the electrocardiogram, echocardiography, Pro BNP, and sST2 values of the patients, as well as any hospitalization, lower respiratory tract infection, organ dysfunction, or need for angiography or surgery during follow-up Data on arrhythmia and death were gathered during a 1-year follow-up. The SPSS software application was used to carry out the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The patients were those with congenital cardiac disease or cardiomyopathy who needed medical care as well as surgical or interventional treatment.

Exclusion Criteria:

* . Excluded from the trial were individuals who had undergone cardiac surgery within past one month, had chronic renal failure, septic shock, myocardial dysfunction related to cardiopulmonary resuscitation, or for whom consent could not be received.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study was conducted in Eskisehir Osmangazi University Pediatric cardiology clinic
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Soluble suppression of tumorigenicity levels with or without major cardiovascular event | baseline
  pg/ml
Pro BNP levels | baseline
  pg/ml
Major cardiovascular event ( such as hospitalization, lower respiratory tract infection, organ dysfunction, or need for angiography or surgery) | 1 year follow up
  rate(%)

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No